CLINICAL TRIAL: NCT05328544
Title: Clinical and Comparative Evaluation of the Results of Autograft Healing of the Tendon of the Semitendinus Muscle in the Tibial Canal, After Reconstruction of the Anterior Cruciate Ligament of the Knee Joint, by the Method of Stabilization of the Screw With a Bioabsorbable Method, With or Without the Use of Autogenous Spongiform Bone Grafts.
Brief Title: Reconstruction of the Anterior Cruciate Ligament of the Knee Joint, by the Method of Stabilization of the Screw With a Bioabsorbable Method, With or Without the Use of Autogenous Spongiform Bone Grafts.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: eMKa MED Medical Center (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-688/2021
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Knee Injuries; Knee Ligament Injury
Keywords: Injury; Rupture; Damage; Reconstruction; Techniques
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Wounds and Injuries; Rupture

STUDY DESIGN:
Intervention Model Description: A- stabilization of the tibial attachment with a bioabsorbable screw (Arthrex) with simultaneous application to the tibial canal of autogenous cancellous bone grafts taken during the drilling of this canal; B- stabilization of the tibial insertion with a bioabsorbable screw (Arthrex) without simultaneous application of autogenous cancellous bone grafts to the tibial canal.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL Reconstruction with the use of autogenous spongiform bone grafts (Experimental): Stabilization of the tibial insertion with a bioabsorbable screw (Arthrex) with simultaneous application to the tibial canal of autogenous cancellous bone grafts taken during the drilling of this canal.
  Interventions: Procedure: ACL reconstruction of the knee joint by arthroscopic technique, with the tibial fixation method using a bioabsorbable screw (Arthrex) with the use of autogenous cancellous bone grafts
- ACL Reconstruction without the use of autogenous spongiform bone grafts (Active Comparator): Stabilization of the tibial attachment with a bioabsorbable screw (Arthrex) without simultaneous application of autogenous cancellous bone grafts to the tibial canal.
  Interventions: Procedure: ACL reconstruction of the knee joint by arthroscopic technique, with the tibial fixation method using a bioabsorbable screw (Arthrex) without the use of autogenous cancellous bone grafts

INTERVENTIONS:
Procedure: ACL reconstruction of the knee joint by arthroscopic technique, with the tibial fixation method using a bioabsorbable screw (Arthrex) with the use of autogenous cancellous bone grafts — Reconstruction of the anterior cruciate ligament (ACL) of the joint the knee stabilization method, a bioabsorbable screw with the use of an autogenous spongy bone graft taken during drilling of the tibial canal into the tibial canate before inserting the screw.
  Arms: ACL Reconstruction with the use of autogenous spongiform bone grafts
Procedure: ACL reconstruction of the knee joint by arthroscopic technique, with the tibial fixation method using a bioabsorbable screw (Arthrex) without the use of autogenous cancellous bone grafts — Reconstruction of the anterior cruciate ligament (ACL) of the joint the knee stabilization method, a bioabsorbable screw without the use of an autogenous spongy bone graft taken during drilling of the tibial canal into the tibial canate before inserting the screw.
  Arms: ACL Reconstruction without the use of autogenous spongiform bone grafts

SUMMARY:
Clinical and comparative evaluation of the results of autograft healing of the tendon of the semitendinus muscle in the tibial canal, after reconstruction of the anterior cruciate ligament of the knee joint, by the method of stabilization of the screw with a bioabsorbable method, with or without the use of autogenous spongiform bone grafts.

DETAILED DESCRIPTION:
Assessment of the results of autograft healing of the tendon of the semitendinus muscle in the tibial canal, after the reconstruction of the anterior cruciate ligament (ACL) of the knee joint using the arthroscopic technique, with the method of tibial stabilization with a bioabsorbable screw (Arthrex) with the use of autogenous transplantation of spongy bone, drilling of the tibial canal inserted into the tibial canal prior to insertion of the screw. The detailed objectives are: comparison of the treatment results - healing and reconstruction of the autograft of the semitendinus tendon in the tibial canal of the knee joint, obtained in the study groups using two methods:

A- stabilization of the tibial attachment with a bioabsorbable screw (Arthrex) with simultaneous application to the tibial canal of autogenous cancellous bone grafts taken during the drilling of this canal and

B- stabilization of the tibial insertion with a bioabsorbable screw (Arthrex) without simultaneous application of autogenous cancellous bone grafts to the tibial canal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Surgery for ACL damage to the knee joint;
* Arthroscopic surgery;
* No prior knee surgical interventions;
* No additional pathologies in this anatomical area;
* Informed consent of the patient to participate in the study.

Exclusion Criteria:

* Age under 18 or over 65;
* Previous surgical interventions in the examined anatomical area;
* Additional pathologies in this area identified as part of preoperative diagnostics;
* Damage to the second knee joint;
* Failure to comply with the rigor of the same rehabilitation treatment protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-08-13 (Estimated); Study Completion 2022-08-13 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | 1 day
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 3 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score (VAS) | 6 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Tegner Activity Scale (TAS) | 1 day
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Scale (TAS) | 3 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Scale (TAS) | 6 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 1 day
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 3 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 6 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
Tegner Lysholm Knee Scoring Scale | 1 day
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale | 3 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale | 6 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Body Mass Index (BMI) | 1 day
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 3 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 6 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Magnetic resonance imaging (MRI) | 6 months after procedure
  1,5 Tesli
Ultrasonography (USG) | 6 months after procedure
  Ultrasound examination on the apparatus with the option of elastometry
Biomechanical examination | 3 months after procedure
  On the Biodex 3 System measuring device
Biomechanical examination | 6 months after procedure
  On the Biodex 3 System measuring device

CONTACTS AND LOCATIONS:
Locations (1):
- eMKa MED Medical Center, Wroclaw, Dolnośląsk, Poland

IPD SHARING:
Plan to Share IPD: No